CLINICAL TRIAL: NCT06263270
Title: A Phase Ia, Multicenter, Double-Blind, Placebo-controlled Study to Evaluate the Safety of CYT-108 for the Therapy of Mild to Moderate Primary Osteoarthritis of the Knee
Brief Title: Evaluation of CYT-108, A Recombinant Protease Inhibitor, for Treatment of Mild To Moderate Primary Osteoarthritis Of The Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytonics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-2023-01
Record Dates: First submitted 2024-01-10; First posted 2024-02-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis
Keywords: arthritis; osteoarthritis; joint pain; joint inflammation; knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis; Arthralgia

STUDY DESIGN:
Intervention Model Description: The Phase 1a trial will be a multicenter, double-blind, randomized, placebo-controlled clinical study to evaluate the safety of two doses of CYT-108 (given at Day 1 and Day 85) in participants with mild to moderate primary OA of the knee, followed out to 26 weeks. A Screening Visit will be performed between twenty-eight days to two days before the first dose, (i.e., Days -28 to -2), and if eligible, participants will attend baseline evaluation on Day 1 to confirm eligibility before randomisation to treatment. The first and second doses will be administered on Day 1 and Day 85 (12 weeks post-first dose, with six follow-up visits on Days 8, 29, 57, 85, 113, and 183; Weeks 1, 4, 8, 12, 16, and 26 weeks post-first dose respectively).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double-blind, placebo-controlled. Neither the investigator, care providers, patients, nor study sponsor have knowledge of the interventions assigned to each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Treatment Arm (CYT-108) (Active Comparator): One intra articular (IA) injection of 5mL at 5mg/mL into one target knee with mild to moderate OA for total of 25mg CYT-108 on Days 1 and 85 (2 injections [50 mg] in total).
  Interventions: Biological: CYT-108, a recombinant protease inhibitor
- Placebo Control Arm (Phosphate Buffered Saline) (Placebo Comparator): Equivalent volume 5mL of phosphate buffer saline, PBS (equal volume to the active treatment arm injection) at the same time intervals as the treatment arm.
  Interventions: Other: Phosphate Buffered Saline (PBS)

INTERVENTIONS:
Biological: CYT-108, a recombinant protease inhibitor — CYT-108 is a recombinant alpha-2-macroglobulin (A2M) variant engineered with increased potency against A Disintegrin and Metalloproteinase with Thrombospondin motifs (ADAMTS) substrates while possessing strong activity against Matrix Metalloproteinases (MMPs) and serine proteases. This A2M variant was engineered with amino acid modifications to the "bait" region (i.e., protease-binding region) of the A2M protein to make the variant at least two fold more effective in inhibiting ADAMTSs compared to wt-A2M without affecting its inhibitory activity toward other proteases (see Investigator Brochure). CYT-108 is not expected to cure osteoarthritis (OA), but it is expected to be the first treatment to slow disease progression by inhibiting cartilage breakdown, resulting in clinically significant outcomes such as pain reduction and improvement in mobility. This hypothesis is supported by our preliminary findings in multiple safety and efficacy studies conducted in rat and canine models of OA.
  Arms: Active Treatment Arm (CYT-108)
Other: Phosphate Buffered Saline (PBS) — Phosphate Buffered Saline (PBS)
  Arms: Placebo Control Arm (Phosphate Buffered Saline)

SUMMARY:
The goal of this Phase 1 study is to investigate the safety of CYT-108, our experimental recombinant protease inhibitor drug candidate for osteoarthritis, in a population of patients suffering from osteoarthritis of the knee. The main questions this study aims to answer are:

1. are two doses of CYT-108, delivered 12 weeks apart, safe when injected directly into the joint?
2. does administration of CYT-108 result in a reduction in pain, stiffness, and improvement in daily physical function?

Participants will either receive a placebo (Phosphate Buffer Saline, PBS) or CYT-108, and will be asked to report their pain/stiffness at weeks 1, 4, 8, 12, 16, and 26 (in a physician's office) after the initial injection, using a questionnaire to be provided by the physician. In addition to reporting the magnitude of pain, participants will also be asked about the onset of pain reduction. Researchers will compare the pain/stiffness scores between the CYT-108-treated to placebo-treated groups along the 26 week duration of the study. Participants will also receive blood draws along the course of the study, and researchers will analyze this blood for the presence of cartilage degradation product in attempt to identify "disease modification" (i.e., a reduction in cartilage degradation) in response to CYT-108 treatment.

DETAILED DESCRIPTION:
The Phase 1a trial will be a multicenter, double-blind, randomized, placebo-controlled clinical study to evaluate the safety of two doses of CYT-108 (given at Day 1 and Day 85) in participants with mild to moderate primary OA of the knee, followed out to 26 weeks. A Screening Visit will be performed between twenty-eight days to two days before the first dose, (i.e., Days -28 to -2), and if eligible, participants will attend baseline evaluation on Day 1 to confirm eligibility before randomization to treatment. The first and second doses will be administered on Day 1 and Day 85 (12 weeks post-first dose, with six follow-up visits on Days 8, 29, 57, 85, 113, and 183 (1, 4, 8, 12, 16, and 26 weeks post-first dose respectively).

At screening, each participant will undergo the informed consent process. After written informed consent is obtained, participants will undergo screening assessments to determine study eligibility. Participants who have not had an X-ray performed within 6 months of screening will undergo an X-ray to determine eligibility. After completing all assessments and meeting study eligibility, the participant will be randomized to receive active treatment or control. Assessments of OA symptoms (WOMAC) will be performed, and blood samples will be obtained at screening and the baseline visit pre-first dose (Day 1) and at specified time-points over the 26-week study period (Weeks 1, 4, 8, 12, 16, and 26).

Approximately twenty-two (22) participants will be randomized in this study in the following manner:

* Participants randomized to Active treatment (12 participants, to assure at least 10 participants to complete the study) will receive one, 5mL (five milliliters) intra-articular injections of CYT-108 (5mg/mL) on each Days 1 and 85, with arthrocentesis prior to injection if clinically appropriate at the time of intervention. Excess fluid in the participant's knee joint will be withdrawn before the drug injection and discarded.
* Participants randomized to Control treatment (10 participants) will receive one, 5mL intra-articular injections of PBS on each Days 1 and 85, with arthrocentesis prior to injection if clinically appropriate at the time of intervention. Excess fluid in the participant's knee joint will be withdrawn before the drug injection and discarded.

Following screening, all participants will have seven site visits on schedule starting with attending the site for the first injection on Day 1, with follow up visits at Weeks 1, 4, 8 and 12. The second injection will be administered at Week 12 after the Investigator has reviewed the participant and confirmed administration of the second dose is acceptable. After this second dose, follow-up evaluations will be conducted in Weeks 16, and 26. At each visit, patients will a combination of physical exams, blood draws, urinalysis, analysis of vital signs, and joint pain/stiffness assessment (using the WOMAC scoring system).

The Week 26 visit will be the end of the study visit (EOS). Participants who withdraw or are withdrawn after the first dose will be asked to attend at early termination visit (ET), at which EOS assessments will be performed. Self-provided rescue medication and any other concomitant medication will be recorded throughout the duration of the study by the study staff or via the participant's diary (ePRO).

ELIGIBILITY:
Inclusion Criteria:

1. Participant with mild to moderate primary knee OA.
2. Provides signed written informed consent before any study procedure is performed.
3. Is willing and able to complete effectiveness and safety questionnaires and can read and understand study instructions.
4. Adult aged 18 years or older at the time of informed consent.
5. Participants of childbearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy test pre-dose on Day 1, and must agree to remain sexually abstinent, or use medically effective contraception (refer to Appendix 14.2) or have a partner who is sterile or same sex, from Screening until at least 3 months after the last treatment. Participants must not be planning to father children or donate sperm from Screening until at least 3 months after the last treatment.
6. Male participants must agree to use a double method of contraception to prevent partner's pregnancy during and 3 months after the last treatment. Male participant should not donate sperm during the same period (for more detail see appendix 14.2).
7. Is ambulatory (assistive devices or knee braces are allowed if used during the study).
8. Has symptomatic OA in the target knee (one knee) either medial or lateral.

   * X-ray confirmation of OA at the target knee prior to screening with a grade 2 or 3 score on the K-L grading scale (Kellgren, 1957) using X-ray performed within 6 months of Screening.
   * Knee pain as demonstrated by an average WOMAC pain scale score of 1.5 - 3 at Screening and pre-dose Day 1.
9. Remains symptomatic despite having received standard of- care therapy, such as daily doses of NSAID or any pain medication leading to the study screening.
10. Has not received corticosteroid injection within 6 weeks prior to screening.
11. Has not received hyaluronic acid treatment, Platelet rich plasma (PRP) or any other protein based or stem cells treatment, or any investigational drug within 12 weeks prior to screening.

Exclusion Criteria:

1. Any of the following:

   1. Grade 4 score on the K-L grading scale for the target knee
   2. Grade 3 score on the K-L grading scale and exhibits at least one Grade 4 characteristic (large osteophytes, marked narrowing of joint space, severe sclerosis, or definite deformity of bone contour)
   3. Acute fracture of the lower limb
   4. Participant with OA in both knees.
2. Medical history of severe bone disease (e.g., osteoporosis, osteonecrosis, joint deformity, instability, or septic arthritis).
3. Has large knee joint effusion, clinically defined as an obvious swelling with loss of the medial sulcus as well as a ballotable patella.
4. Has another disease that can affect the health of the knee (e.g., chronic hemochromatosis; sickle cell anemia; arthropathies of systemic diseases such as chondrocalcinosis, gout, pseudogout, psoriasis, hemophilia, and infectious diseases of the joints).
5. Significant joint infection in the target knee or inflammation or skin disorder in the injection area of the target knee.
6. Fibromyalgia, anserine bursitis, lumbar radiculopathy, neurogenic or vascular claudication, vascular insufficiency of lower limbs, or peripheral neuropathy.
7. Patella femoral instability.
8. History of cartilage allograft, autograft or microfracture in the study knee.
9. Has diseases that may interfere:

   1. Severe infectious disease with or without fever. COVID-19 patients will not be permitted until two negative tests are produced.
   2. The history of suffering from migraine headache and requires ongoing pain medications that are prohibited per protocol.
   3. Any significant chronic skin disorders, active skin or soft tissue infection that could interfere with the evaluation of the injection site.
   4. Malalignment/deformity of the leg
   5. Active Chronic Obstructive Pulmonary Disease (COPD) or Asthma that may require periodic treatment with steroids during the study period.
   6. Active malignancy receiving treatment, or prior history of any malignancy, except for basal cell carcinoma or squamous cell carcinoma of the skin treated at least 1 year before screening.
10. Psychiatric, neurological disorders, or cognitive impairment severe enough that the individual is unable to provide informed consent, in the judgement of the Investigator.
11. Incarcerated or confined.
12. Has medical-legal, personal injury, ongoing litigation, or a worker's compensation claim(s).
13. Smokers, tobacco users and any nicotine administration through vaping or patches.
14. History of alcohol or drug abuse.
15. Received corticosteroid injection for any indication within 6 weeks prior to screening.
16. Pregnant and breast-feeding participants or planning to get pregnant during and 6 months after the study is completed.
17. Clinically significant abnormal screening laboratory results (other than those related to OA)
18. Clinically significant abnormal vital signs or physical examination findings (other than those related to OA).
19. Received hyaluronic acid treatment, Platelet rich plasma (PRP) or any other protein based or stem cells treatment, or any investigational drug within 12 weeks prior to screening.
20. Any condition that, in the opinion of the Clinical Investigator, might interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Day 0; Weeks 1, 4, 8, 12, 16, 26
  Frequency and severity of Adverse Events (AE), Serious Adverse, Events (SAE) and Treatment-Emergent Adverse Events (TEAEs).
Blood Pressure | Day 0; Weeks 1, 4, 8, 12, 16, 26
  Systolic and Diastolic blood pressure [mmHg]
Heart Rate | Day 0; Weeks 1, 4, 8, 12, 16, 26
  Heart rate [beats per minute]
Respiratory Rate | Day 0; Weeks 1, 4, 8, 12, 16, 26
  Respiratory rate [breaths per minute]
Body Temperature | Day 0; Weeks 1, 4, 8, 12, 16, 26
  Body temperature [°C]
Titer of Human Anti-Drug Antibody | Day 0; Weeks 1, 4, 8, 12, 16, 26
  Change from baseline in human anti-drug antibody (HADA) to evaluate the immune response toward the new bait region of the molecule (assay to be developed).

SECONDARY OUTCOMES:
Change in WOMAC Scores (Pain, Stiffness, and Difficulty Performing Daily Activities) | Day 0; Weeks 1, 4, 8, 12, 16, 26
  Changes in pain, stiffness, and difficultly in performing daily activities in the treatment group will be compared to the control group using participant's own assessment at 1, 4, 8, 12, 16, and 26 weeks after first intra-articular injection of CYT-108 into the target knee, as determined by the Western Ontario and McMaster Universities Osteoarthritis Index NRS 3.1 (WOMAC). The WOMAC is divided into three subscales: WOMAC-A (pain, 5 questions, 0-10), WOMAC-B (stiffness, 2 questions, 0-10), and WOMAC-C (daily physical function, 17 questions, 0-10). The WOMAC total score ranges from 0-240, where a higher score indicates a worse outcome.
Time of Onset | Day 0; Weeks 1, 4, 8, 12, 16, 26
  Time of onset of pain determined by asking enrolled participants whether they are aware of the onset of meaningful pain reduction and the time it took for the pain reduction

OTHER OUTCOMES:
Concentration of Cartilage Degradation Fragments in Blood Plasma | Day 0; Weeks 1, 4, 8, 12, 16, 26
  Aggrecan fragment neoepitope (ARGS) concentration in blood plasma, as a biomarker for disease modification (e.g., attenuation of cartilage breakdown), in the treatment group will be compared to the control group using a commercially available ELISA assay at 1, 4, 8, 12, 16, and 26 weeks after first intra-articular injection of CYT-108 into the target knee.

CONTACTS AND LOCATIONS:
Overall Officials: Joey Bose, MS, Study Director — Cytonics Corporation; Lewis Hanna, PhD, Study Director — Cytonics Corporation; Gaetano Scuderi, MD, Study Director — Cytonics Corporation
Locations (3):
- Australia (3):
  - University of Sunshine Coast Clinical Trials, Sunshine Coast, Birtinya QLD
  - Novatrials, Kotara, New South Wales
  - Emeritus Research, Camberwell, Victoria

IPD SHARING:
Plan to Share IPD: No